CLINICAL TRIAL: NCT02556905
Title: REVLIMID® Drug Use Examination
Brief Title: A Study to Collect and Evaluate the Safety and Efficacy Information of Korean Multiple Myeloma Patients Treated With REVLIMID®, After Approval of Marketing Authorization for New Drug in Korea
Status: Completed | Type: Observational
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: NIPMS-RV-KR-001
Record Dates: First submitted 2015-09-21; First posted 2015-09-22 (Estimated); Last update posted 2017-12-04 (Actual); Status verified 2017-11

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Revlimid; Lenalidomide; Observational; Korea; Post Marketing Surveillance[PMS]
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide; Dexamethasone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Korean patients: All Korean patients intended to be treated with REVLIMID® according to the approved package insert
  Interventions: Drug: REVLIMID®; Drug: Dexamethasone

INTERVENTIONS:
Drug: REVLIMID® — The recommended starting dose of REVLIMID® is 25mg/day with water orally administered as a single 25mg capsule on Days 1-21 of repeated 28-day cycles. Dose can be adjusted upon the clinical laboratory result.
Drug: Dexamethasone — The recommended dose of dexamethasone is 40mg/day on Days 1-4, 9-12, and 17-20 of each 28-day cycle for the 4 cycle of therapy and then 40mg/day orally on Days 1-4 every 28 days.

SUMMARY:
The main purpose of REVLIMID® DUE (Drug Use Examination) is to collect and evaluate the safety information of Korean Multiple Myeloma patients treated with REVLIMID® according to the approved package insert, after approval of marketing authorization for new drug in Korea. In addition, the efficacy information of REVLIMID® in clinical practice is collected and evaluated. This DUE is a multi-centre, observational and non-interventional post-marketing surveillance.

The patients can be recruited through both Drug Use Examination after the initiation of Post Marketing Surveillance(contract with institution) and Patient Access Program(PAP) that was performed before REVLIMID® reimbursement.

Total 624 patient has enrolled in PMS by 07Sep2016. Validation process for eligibility for safety assessment has been conducted by site monitoring process by 07Dec2016.

REVLIMID® DUE is to investigate frequency and change of Adverse Events(AEs) /Adverse Drug Reactions(ADRs), Serious Adverse Events(SAEs)/Serious Adverse Drug Reactions(SADRs), unexpected AE/ADR and unexpected SAE/SADR, and to scrutinize factors influencing safety & efficacy of the drug.

It is necessary to examine patients' demographics and baseline characteristics, medical history, status of REVLIMID® treatment, concomitant medication and evaluation of safety and final efficacy (best response) assessment.

ELIGIBILITY:
Inclusion Criteria:

* Korean male or female who are diagnosed with Multiple Myeloma
* In-patients or out patients during the REVLIMID® Drug Use Examination period who are intended to be treated with REVLIMID ®
* Patients who are registered for Risk Management Program of Celgene

Exclusion Criteria:

* There's no exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All Korean patients who are intended to be treated with REVLIMID® and must be registered in risk management program according to the approved package insert.
Sampling Method: Non-Probability Sample
Enrollment: 624 (Actual)
Dates: Start 2011-03-09 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
Adverse events (AEs) | Up to 6 years
  Number of participants with adverse events

SECONDARY OUTCOMES:
Overall response rate | Up to 6 years
  Number of participants with response based on International Myeloma Working Group Criteria for Multiple Myeloma

CONTACTS AND LOCATIONS:
Overall Officials: Miran Moon, Study Director — Celgene Korea
Locations (25):
- South Korea (25):
  - Hallym University Sacred Heart Hospital, Anyang
  - Soon Chun Hyang University Hospital Bucheon, Bucheon-si
  - Inje University Busan Paik Hospital, Busan
  - Inje University Haeundae Paik Hospital, Busan
  - Dong-a University Medical Center, Busan
  - Pusan National University Hospital, Busan
  - Kosin University Gospel Hospital, Busan
  - Kyungpook National University Hospital, Daegu
  - Chungnam National University Hospital, Daejeon
  - Hwasun Chonnam National University Hospital, Hwasun-gun
  - Chonbuk National University Hospital, Jeonju
  - Inje University Sanggye Paik Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Konkuk University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - Boramae Medical Center, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Ulsan University Hospital, Ulsan
  - Wonju Severance Christian Hospital, Wŏnju
  - Pusan National University Yangsan Hospital, Yangsan